CLINICAL TRIAL: NCT03607513
Title: A Double-blind, Placebo-controlled, Randomized, Single and Multiple Ascending Dose Study to Investigate the Safety, Tolerability, and Pharmacokinetics of JNJ-64264681 in Healthy Male and Female Subjects
Brief Title: A Study to Investigate the Safety, Tolerability, and Pharmacokinetics of JNJ-64264681 in Healthy Male and Female Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: CR108457; 2018-000428-32 (EudraCT Number); 64264681EDI1003 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2018-07-24; First posted 2018-07-31 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — JNJ-64264681

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single Ascending Dose (SAD) (Experimental): The SAD part will consist of 6 escalating dose cohorts and 1 fed cohort of healthy male participants, 2 dose escalating cohorts of healthy female participants, and 1 solid dose formulation (capsule) cohort of healthy male participants, who will be dosed after completion of the dose escalation cohorts. Participants in each cohort (except for the solid dose formulation cohort) will receive JNJ-64264681 or Placebo on Day 1, orally. In the solid dose formulation cohort, participants will receive JNJ-64264681 capsule on Day 1. Doses for the female cohorts and fed cohort will be selected based on safety, tolerability, pharmacokinetics (PK),and pharmacodynamic (PD) data from preceding cohorts and the dose for the solid dose formulation cohort will be selected and approximately equal to a dose previously studied in the single ascending dose cohorts.
  Interventions: Drug: JNJ-64264681; Drug: Placebo
- Multiple Ascending Dose (MAD) (Experimental): The MAD part will consist of 3 dose escalation cohorts of males and females. Participants will receive once-daily oral doses of JNJ-64264681 or placebo for 10 consecutive days.
  Interventions: Drug: JNJ-64264681; Drug: Placebo

INTERVENTIONS:
Drug: JNJ-64264681 — For all cohorts except the solid dose formulation cohort, JNJ-64264681 wlll be administered as oral solution. For the solid dose formulation cohort, JNJ-64264681 will be provided as capsules for oral administration.
Drug: Placebo — Matching placebo to JNJ-64264681 will be administered as oral solution.

SUMMARY:
The primary purpose of this study is to investigate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of JNJ-64264681 in healthy participants after single and multiple oral doses.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have a body mass index (BMI) between 18.0 and 30.0 kilogram per meter square (kg/m^2) (BMI = weight[kg]/height[m]^2), and a body weight of not less than 50 kilogram (kg)
* Participant must be healthy on the basis of physical examination, medical history, vital signs, and 12-lead Electrocardiogram (ECG) performed at screening and Day -1
* Participant must be healthy on the basis of clinical laboratory tests performed at screening and Day -1. If the results of the serum chemistry panel, coagulation, hematology, or urinalysis are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant. This determination must be recorded in the participant's source documents and initialed by the investigator
* Participant must sign an informed consent form (ICF) indicating that he or she understands the purpose of, and procedures required for, the study and is willing to participate in the study
* Female participants must not be of childbearing potential by fulfilling 1 of the criteria below: a) Be over 45 years of age with no menses for 12 months without an alternative medical cause, with screening follicle stimulating hormone (FSH) levels of greater than (>)40 International Units Per Liter (IU/L) or milli-international units per milliliter (mIU/mL). b) Be permanently surgically sterile. Permanent surgical sterilization methods include hysterectomy, bilateral salpingectomy, bilateral tubal occlusion/ligation procedures, and bilateral oophorectomy. Documentation of FSH levels is not required in the case of surgical sterility

Exclusion Criteria:

* Participant has current, or history of clinically significant medical illness including, but not limited to, liver or renal insufficiency, significant cardiac (including heart valve disease), vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances
* Participant has a history of abnormal bleeding or bruising
* Participant has a history of atrial fibrillation or history of arrhythmias
* Participant has history of malignancy within 5 years before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy, which in the opinion of the investigator, with concurrence with the sponsor's medical monitor, is considered cured with minimal risk of recurrence)
* Participant has known allergies, hypersensitivity, or intolerance to polyethylene glycol 400 (PEG400) (vehicle for JNJ-64264681 for oral solution dosing) for participant in a cohort where study drug is to be dosed as an oral solution, or to microcrystalline cellulose, lactose monohydrate, croscarmellose sodium, silica dioxide, sodium lauryl sulfate, magnesium stearate, or gelatin (excipients in the solid dose formulation (capsule) of JNJ-64264681) for participant in a solid dose formulation cohort

Ages: 18 Years to 58 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2019-08-09 (Actual); Study Completion 2019-08-09 (Actual)

PRIMARY OUTCOMES:
Single Ascending Dose (SAD): Number of Participants with Adverse Events | Up to Day 14
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Multiple Ascending Dose (MAD): Number of Participants with Adverse Events | Up to Day 24
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
SAD: Maximum Observed Plasma Concentration (Cmax) | Up to Day 4
  Cmax is the maximum observed plasma JNJ-64264681 concentration.
MAD: Maximum Observed Plasma Concentration (Cmax) | Up to Day 13
  Cmax is the maximum observed plasma JNJ-64264681 concentration.
SAD: Time to Reach Maximum Observed Plasma Concentration (Tmax) | Up to Day 4
  Tmax is defined as actual sampling time to reach maximum observed concentration.
MAD: Time to Reach Maximum Observed Plasma Concentration (Tmax) | Up to Day 13
  Tmax is defined as actual sampling time to reach maximum observed concentration.
SAD: Time to Last Quantifiable Plasma Concentration (Tlast) | Up to Day 4
  The Tlast is the time to last observed quantifiable plasma concentration.
MAD: Time to Last Quantifiable Plasma Concentration (Tlast) | Up to Day 13
  The Tlast is the time to last observed quantifiable plasma concentration.
SAD: Area Under the Plasma Concentration-time Curve From Time Zero to 24 Hours (AUC[0-24]) | Day 1: Up to 24 hours post-dose
  AUC (0-24) is the area under the plasma concentration-time curve from time zero to 24 hours.
MAD: Area Under the Plasma Concentration-time Curve From Time Zero to 24 Hours (AUC[0-24]) | Day 1: Up to 24 hours post-dose
  AUC (0-24) is the area under the plasma concentration-time curve from time zero to 24 hours.
SAD: Area Under the Plasma Concentration-time Curve From Time 0 to Time of the Last Observed Quantifiable Concentration (AUClast) | Up to Day 4
  AUClast is defined as area under the plasma JNJ-64264681 concentration-time curve from time 0 to time of the last observed quantifiable concentration.
MAD: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) | Day 10
  AUCtau is area under the plasma JNJ-64264681 concentration-time curve during a dosing interval (tau) at steady-state.
SAD: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) | Up to Day 3
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z); wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.
SAD: Apparent Elimination Half-life (t1/2) | Up to Day 3
  t1/2 is apparent elimination half-life of JNJ-64264681 associated with the terminal slope (z) of the semi-logarithmic drug concentration-time curve.
MAD: Apparent Elimination Half-life (t1/2) | Up to Day 13
  t1/2 is apparent elimination half-life of JNJ-64264681 associated with the terminal slope (z) of the semi-logarithmic drug concentration-time curve.
MAD: Accumulation Ratio | Up to Day 13
  MAD: Accumulation Ratio obtained by dividing AUC of JNJ-64264681 at two different time points.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Clinical Pharmacology Unit, Merksem, Belgium